CLINICAL TRIAL: NCT00069420
Title: Cognitive-Motivational Behavior Therapy for Gamblers
Brief Title: Cognitive Motivational Behavior Therapy for Gamblers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University at Albany (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Edelgard Wulfert, Dean, College of Arts & Sciences, University at Albany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R21MH064568 (NIH); R21MH064568 (NIH); DSIR AT-AS
Record Dates: First submitted 2003-09-24; First posted 2003-09-25 (Estimated); Last update posted 2014-01-01 (Estimated); Status verified 2013-12

CONDITIONS: Gambling
MeSH Terms: conditions — Gambling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Cognitive Motivational Behavior Therapy

SUMMARY:
This study will evaluate the effectiveness of cognitive motivational behavior therapy (CMBT) in treating pathological gamblers.

DETAILED DESCRIPTION:
Pathological gambling is developing into a serious public health problem. The rise in gambling problems has stimulated treatment studies, but little progress has been made. A particular concern is the high dropout rates from treatment studies; gamblers often seek treatment, but fail to complete it and relapse. This study will test the effectiveness of CMBT in helping to increase retention rates in gambling treatment studies.

The first step in this study is designed to enhance gamblers' readiness for change. When participants are committed to change, CMBT will then address specific cognitive biases regarding the notion of randomness, which is thought to lie at the heart of gambling problems. Behavioral components will also be used to enhance gamblers' coping skills.

The participants in this study will be randomly assigned to either CMBT or a Gambler's Anonymous control group. Participants will be assessed prior to and after treatment and at 3- and 6-month follow-up visits. Interviews and questionnaires will be used to assess participants.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV criteria for pathological gambling
* Eighth grade reading ability
* Reside in the Albany, NY area

Exclusion Criteria:

* Diagnosis of serious psychopathology, including psychosis, bipolar disorder, or alcohol or other substance dependence

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40
Dates: Start 2003-09; Primary Completion 2007-01 (Actual); Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University at Albany - SUNY, Albany, New York, United States